CLINICAL TRIAL: NCT01394068
Title: SICS: A Prospective, Non-randomized Observational Trial of Selenium in Cardiac Surgery
Brief Title: Prospective, Non-randomized Observational Trial of Selenium in Cardiac Surgery
Acronym: SICS
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: PI: PD Dr. Steffen Rex, Clinic for Anaesthesiolgy; Clinical Trial Center Aachen
Other Study IDs: CTC-A 10-013 SICS
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Selenium Deficiency
Keywords: Selenium level; Various blood values; Duration of artificial respiration; Residence in ICU/ Hospital; SOFA-Score; SAPS-Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Procalcitonin, CRP, IL-6, IL-10, Leukocytes, Thrombocytes, Bilirubin, Creatinine, Lactate, Albumin, AT-III
Oversight: Data Monitoring Committee: No

SUMMARY:
In this observational study the effect of selenium supplementation on the postoperative inflammatory response and clinical course should be examined in (approximately 100) adult patients undergoing elective heart surgery combined with extracorporeal circulation.

Selenium is one of the essential trace elements with a variety of important immunological and antioxidant properties. The pathophysiological relevance of different selenium-dependent reactions has already been demonstrated in human and in animal experiments. It is essential for the enzymatic functions of selenium-containing proteins such as the glutathione peroxidase, which in turn affects the leukotriene, thromboxane and prostacyclin metabolism. In addition, selenium has a significant influence on various liver enzymes, therefore selenium deficiency leads to oxidative or chemically induced liver damage.

DETAILED DESCRIPTION:
Heart Surgery on the heart-lung machine involves, inter alia, by ischemia and reperfusion, the release of reactive oxygen radicals and nitrogen oxide (NO), which damage DNA after reaction with peroxynitrite, and Lipid-/Endothelmembrane Protein. The formation and consumption of peroxynitrite can be reduced by intake of sodium selenite and the subsequent formation of selenoprotein P. Since there is no storage for selenium, but the synthesis of selenium-dependent enzymes is regulated by selenium resorption, the supplementation of selenium is a potentially useful application in patients undergoing cardiac surgery.

After induction of anaesthesia and before connecting to the heart-lung machine the patients get applied 2000μg sodium selenite (Selenase® T pro injection) intravenously (as a bolus infusion over 30 minutes).

Furthermore, they get infused 1000μg sodium-selenite on each ICU-treatment day (also about 30 minutes). In addition, various blood values are recorded daily (including selenium levels) within the routine blood samples. As the collection of these parameters is necessary anyway, it constitutes no additional burden on the patient. Shortly before the transfer to general ward there will be a final clinical examination.

In case of selenium level of 170μg per liter whole blood the employee of the laboratory immediately informs the investigator by fax and requests a new blood sample for control purposes (reference value for selenium in whole blood according to product information 100-144µg/ l). As long as the selenium level of the second sample is not higher than 230μg selenium per liter whole blood, there are no further precautions necessary according to the manufacturer's recommendations. In case of selenium level above 230μg /l, the investigator will be informed by fax without delay and the donation of investigational product will be interrupted immediately. If a patient shows clinical signs of selenium toxicity (garlic-like breath odor, fatigue, nausea, diarrhea, abdominal pain) it occurs an immediate termination of the selenium dose, initiating symptomatic counteractive measures and further control samples.

All blood samples are taken by vascular catheters, which are already set for surgery or for intensive care treatment, independent of the observational study.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Elective heart surgery on the heart-lung-machine
* Written informed consent
* Inclusion into observational study at the latest on the last evening before surgery

Exclusion Criteria:

* Patients not capable of consenting
* pregnant women or women of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 adult patients (male and female), capable of consenting, undergoing elective cardiac surgery on the heart-lung-machine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aachen, Aachen, Germany